CLINICAL TRIAL: NCT00605540
Title: Three-years Follow-up of Diagnostic and Prognostic Markers in Chronic Obstructive Pulmonary Disease
Brief Title: Chronic Obstructive Pulmonary Disease Markers and Prognosis
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Irma de Godoy, PhD, UPECLIN HC FM Botucatu Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-06
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Survival; Exacerbation; Disease markers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study COPD population: Patients with diagnosis of mild to very severe chronic obstructive pulmonary disease

SUMMARY:
The study aim is to verify the association between the changes in markers of disease and patient´s prognosis in chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
In a previous study, 133 COPD patients were followed-up during the period of one-year. Analyses of the association between baseline characteristic and the occurence of disease exacerbation was performed. In this study, the patients included in the previous research will be contacted and invited to participate in a complete evaluation after a three-year period. The association of the changes in dyspnea perception, spirometry variables, body composition, quality of life and exercise tolerance measures with disease prognostic will be studied.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to the GOLD criteria

Exclusion Criteria:

* Asthma
* Inability to perform pulmonary function and exercise tolerance tests
* Recent myocardial infarction or unstable angina
* Congestive heart failure: class III/IV

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irma de Godoy, PhD, MD, Study Chair — Botucatu School of Medicine
Locations (1):
- Botucatu School of Medicine, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] Ferrari R, Tanni SE, Caram LM, Correa C, Correa CR, Godoy I. Three-year follow-up of Interleukin 6 and C-reactive protein in chronic obstructive pulmonary disease. Respir Res. 2013 Feb 20;14(1):24. doi: 10.1186/1465-9921-14-24. PMID 23425215
- [Derived] Ferrari R, Tanni SE, Caram LM, Naves CR, Godoy I. Predictors of health status do not change over three-year periods and exacerbation makes difference in chronic obstructive pulmonary disease. Health Qual Life Outcomes. 2011 Dec 9;9:112. doi: 10.1186/1477-7525-9-112. PMID 22152155

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Obstructive Pulmonary Disease Markers Over Three Years: All patients were evaluated at baseline and attended at the clinics every six months for three years or until death.
Period: Overall Study
Arm/Group | Chronic Obstructive Pulmonary Disease Markers Over Three Years
Started | 133
Completed | 95
Not Completed | 38
Not completed — Death | 15
Not completed — Lost to Follow-up | 23

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Obstructive Pulmonary Disease Markers Over Three Years
Number analyzed (Participants) | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 92
Region of Enrollment [Number; unit: participants]
  Brazil | 133

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in the First Second (FEV1)
Description: FEV1 values were measured by Spirometry using the KOKO Spirometer, before and 15 minutes after the inhalation of 400mcg of salbutamol.
Time Frame: Baseline and after three years
Population: The sampling frame for this study was consecutive COPD patients recruited from the outpatient clinic of Botucatu Medical School.
Measure: Median (Inter-Quartile Range); unit: Percentage predicted
Arm/Group | Chronic Obstructive Pulmonary Disease Markers Over Three Years
Number analyzed (Participants) | 95
Percentage predicted
  Baseline assessment | 54 [41 to 73]
  After three-year assessment | 54 [40 to 70]
Statistical Analysis 1: Comparison: Chronic Obstructive Pulmonary Disease Markers Over Three Years; All data were analyzed using SigmaStat 3.2 (Inc., USA) software. Mean ± SD or median interquartile range (25-75%) was used depending on the data distribution. Wilcoxon test was applied to compare the characteristics at baseline to those observed after 3 years; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Exercise Tolerance
Description: Tolerance exercise was evaluated by six-minute walking distance(6MWD)according to the American Thoracic Society guidelines.Patients were instructed to walk, attempting to cover as much ground as possible within 6 min. A research assistant timed the walk, and standardized verbal encouragement was given.
Time Frame: Baseline and after three years
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Chronic Obstructive Pulmonary Disease Markers Over Three Years
Number analyzed (Participants) | 95
meters
  Baseline assessment | 438 (86)
  After three-year assessment | 412 (100)

3. Primary Outcome: Body Composition
Description: Body composition was evaluated by Body Mass Index (BMI), which is dividing weight in kilograms by height in square meters.
Time Frame: Baseline and after three years
Measure: Median (Inter-Quartile Range); unit: Kg/m^2
Arm/Group | Chronic Obstructive Pulmonary Disease Markers Over Three Years
Number analyzed (Participants) | 95
Kg/m^2
  Baseline assessment | 25 [22 to 29]
  After three-year assessment | 25 [22 to 29]

4. Primary Outcome: Dyspnea
Description: Dyspnea was evaluated by Medical Research Council scale (MRC). MRC scale consists of only five items and it is based on activities that cause dyspnea. The patient reports the degree of dyspnea by choosing a value between 1 and 5. A higher number indicates greater sensation of dyspnea.
Time Frame: Baseline and after three years
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Chronic Obstructive Pulmonary Disease Markers Over Three Years
Number analyzed (Participants) | 95
Scores on a scale
  Baseline assessment | 1 [1 to 2]
  After three-year assessment | 2 [1 to 3]

5. Primary Outcome: Health Status
Description: Saint George's Respiratory Questionnaire (SGRQ)was used to evaluate patient's health status. SGRQ includes three domains: symptoms, activities and impact of the disease. Each domain has a minimum score (zero) and maximum (662.5, 1209.1, and 2117.8, respectively). A total score is also calculated based on the results of three domains, with a score maximum of 3989.4. The total score is referred to as the percentage achieved by the patient related to this maximum score. Minimum score means there is no impairment in the health status and high score means maximum dysfunction.
Time Frame: Baseline and after three years
Measure: Mean (Standard Deviation); unit: Percentage of total score
Arm/Group | Chronic Obstructive Pulmonary Disease Markers Over Three Years
Number analyzed (Participants) | 95
Percentage of total score
  Baseline assessment | 42 (19)
  After three-year assessment | 44 (19)

ADVERSE EVENTS:
Arm/Group | Chronic Obstructive Pulmonary Disease
Serious Adverse Events (participants affected / at risk) | 0/133
Other Adverse Events (participants affected / at risk) | 0/133

LIMITATIONS AND CAVEATS:
We excluded patients with comorbidities; therefore, many patients seen in clinical practice may not have been well represented in our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No